CLINICAL TRIAL: NCT05037123
Title: Optimizing the Use of Ketamine to Reduce Chronic Postsurgical Pain
Acronym: KALPAS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 21-00715
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Chronic Postsurgical Pain
Keywords: Mastectomy; Post-Mastectomy; Ketamine
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, study members, and treating clinicians will be blinded to intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm 1 Continuous ketamine infusion group (Active Comparator): Continuous ketamine infusion (0.35 mg/kg after induction, followed by 0.25 mg/kg/hr until 2 hours after surgery) plus saline IV dose in post-anesthesia care unit
  Interventions: Drug: Continuous ketamine infusion
- Arm 2 Ketamine + Saline group (Active Comparator): Saline dose and infusion intraoperatively, then single-dose IV ketamine (0.60 mg/kg) in post-anesthesia care unit plus 2 hours of saline administration after surgery
  Interventions: Drug: Ketamine + Saline
- Arm 3 Placebo group (Placebo Comparator): Placebo, Saline dose and infusion intraoperatively, then saline IV dose in post-anesthesia care unit plus 2 hours of saline administration after surgery
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Continuous ketamine infusion — Continuous ketamine infusion (0.35 mg/kg after induction, followed by 0.25 mg/kg/hr until 2 hours after surgery) plus saline IV dose in post-anesthesia care unit
  Arms: Arm 1 Continuous ketamine infusion group
Drug: Ketamine + Saline — Saline dose and infusion intraoperatively, then single-dose IV ketamine (0.60 mg/kg) in post-anesthesia care unit plus 2 hours of saline administration after surgery
  Arms: Arm 2 Ketamine + Saline group
Other: Placebo — Placebo, Saline dose and infusion intraoperatively, then saline IV dose in post-anesthesia care unit plus 2 hours of saline administration after surgery
  Arms: Arm 3 Placebo group

SUMMARY:
The study utilizes a 3-arm placebo-controlled RCT to study the effectiveness of ketamine in reducing chronic post-mastectomy pain. Participants randomized to the first arm will receive a 0.35 mg/kg dose after induction, followed by a 0.25 mg/kg/hr infusion during surgery (up to a maximum of 6 hours) and continued for 2 hours postoperatively. Participants in the second arm will receive a single dose of 0.6 mg/kg of ketamine in the post-anesthesia care unit, and the final group will serve as the control group and receive saline (no ketamine).

DETAILED DESCRIPTION:
This is a phase 3, multicenter, randomized, double-blind, placebo-controlled trial to study the effectiveness of ketamine in reducing PMPS. In a 3-arm, parallel-group study, approximately 750 adult women undergoing mastectomy or prophylactic mastectomy for oncologic reasons will be randomized to one of three arms. Participants in the first arm will receive continuous ketamine infusion starting after anesthetic induction (0.35 mg/kg dose after induction, followed by a 0.25 mg/kg/hr infusion during surgery (with a maximum infusion of 6 hours) plus a postoperative saline dose, and continuation of 0.25 mg/kg/hr ketamine infusion for 2 hours postoperatively). Participants in the second arm will receive a dose of saline after induction, followed by a saline infusion during the surgery plus a single dose of 0.6 mg/kg of ketamine in the PACU, and 2 hours of saline infusion after surgery. The final group will serve as the control group and receive an intraoperative dose of saline, followed by saline infusion plus a postoperative saline dose and 2 hours of saline infusion after surgery. Participants will be followed at 1 and 7 days and 1, 3, 6, and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Woman 18 years of age or older
* Undergoing elective breast surgery for oncologic indication as follows: unilateral or bilateral mastectomy, prophylacticmastectomy, +/- lymph node dissection, +/- immediate or delayed reconstruction.
* No distant metastases

Exclusion Criteria:

* History of cognitive impairment or clinical signs of altered mental status (AMS) that may interfere with adherence to study procedures and/or participant safety. Clinical signs of AMS may include but are not limited to: confusion, amnesia, disorientation, fluctuating levels of alertness, etc.
* Past ketamine or phencyclidine misuse or abuse
* Schizophrenia or history of psychosis
* History of post-traumatic stress disorder
* Known sensitivity or allergy to ketamine
* Liver or renal insufficiency
* History of uncontrolled hypertension, chest pain, cardiac arrhythmia, stroke, head trauma, intracranial mass or hemorrhage, glaucoma, porphyria, uncontrolled thyroid disease, or other contraindication to ketamine
* Lamotrigine, alfentanil, physostigmine, or 4-aminopyridine use
* Currently Pregnant
* Body mass index (BMI) equal to or greater than 41
* Non-English or non-Spanish speaker
* Currently participating in another pain interventional trial
* Unwilling to comply with all study procedures and be available for the duration of the study
* Patient is American Society of Anesthesiologists (ASA) physical status 4, 5, or 6
* Patient has started or undergone hormone therapy for gender transition into male.
* Patient scheduled for any bilateral (or greater) flap reconstruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 765 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
BPI pain severity subscale score | 3 months
  The Brief Pain Inventory short form (BPI) pain severity subscale assesses pain at its worst, least, average, and current in the past 24 hours.
  The score ranges from 0 to 10 for each item. The average of the four items will be used. The BPI scale defines pain as follows: Worst Pain Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain.

SECONDARY OUTCOMES:
BPI pain severity and pain interference subscales score | Baseline, 1 and 7 days and 1, 3*, 6, and 12 months after surgery
  BPI assesses pain severity and interference. The interference subscale measures how much pain has interfered with general activities such as walking and working. Additionally, it inquires about interference in mood, enjoyment of life, relationships, and sleep. The BPI scale defines pain as follows: Worst Pain Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain.
Incidence of PMS: BPI average pain score | Baseline, 3, 6, and 12 months after surgery
  The BPI pain severity subscale assesses pain at its worst, least, average, and current in the past 24 hours.
  We will use participant's average pain item to assess incidence of PMPS. A score greater than 3 (0-10 scale) will be considered clinically meaningful chronic pain.
Pain in the surgical site (chest wall, axilla, and/or arm): BCPQ Score | 7 days and 1, 3, 6, and 12 months after surgery
  The Breast Cancer Pain Questionnaire (BCPQ) assesses pain location, frequency, and severity as well as sensory disturbance after breast surgery. The BCPQ queries patients about pain severity (scores 1-10) and frequency (scores 5 [constantly], 4 [daily], 3 [occasionally], 2 [weekly], 1 [monthly], and 0 [never]) in four surgically related body areas (breast, axilla, chest wall, arm).
PROMIS Depression and Anxiety Short Form Scores | Baseline, 7 days and 1, 3, 6, and 12 months after surgery
  Anxiety and depressive symptoms are prevalent in patients undergoing surgery for breast cancer and are risk factors for PMPS. The PROMIS assessments are designed to measure anxiety and depression symptoms. Each assessment will generate a raw score based on participant-reported answers, where the raw score is then converted into a t-score ranging from 0-100; higher scores indicate greater symptoms of anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, MD, PhD, Principal Investigator — NYU Langone Health; Lisa Doan, MD, Principal Investigator — NYU Langone Health
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas, Little Rock, Arkansas
  - Rush University Medical Center, Chicago, Illinois
  - Brigham and Women's Hospital - Harvard University, Chestnut Hill, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University at St. Louis Medical Center, St Louis, Missouri
  - NYU Langone Health (Tisch Hospital, Kimmel Pavilion), New York, New York
  - New York Presbyterian Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center - Albert Einstein College of Medicine, The Bronx, New York
  - University of Pittsburgh - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - University of Texas - Southwestern Medical Center, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to the PI. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to Jing.Wang2@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Wang J, Doan LV, Axelrod D, Rotrosen J, Wang B, Park HG, Edwards RR, Curatolo M, Jackman C, Perez R; NCATS Trial Innovation Network. Optimizing the use of ketamine to reduce chronic postsurgical pain in women undergoing mastectomy for oncologic indication: study protocol for the KALPAS multicenter randomized controlled trial. Trials. 2024 Jan 19;25(1):67. doi: 10.1186/s13063-023-07884-y. PMID 38243266

DOCUMENTS (1):
  • Informed Consent Form (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT05037123/ICF_000.pdf